CLINICAL TRIAL: NCT00133107
Title: A Single Center, Open-label, Pilot Study Evaluating the Safety and Effectiveness of Subcutaneous Efalizumab in the Treatment of Oral Lichen Planus
Brief Title: Safety and Effectiveness of Efalizumab to Treat Oral Lichen Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Michael P.Heffernan, MD, Washington University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP-efalizumab
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-08

CONDITIONS: Lichen Planus, Oral
MeSH Terms: conditions — Lichen Planus, Oral | interventions — efalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: efalizumab

SUMMARY:
This study is to determine whether efalizumab 1.0mg/kg given by subcutaneous injection for 12 weeks is effective in treating oral lichen planus.

This is a 20 week, single center, open-label pilot study to enroll 5 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Subject able and willing to comply with study requirements for the full duration of the study.
* Age > 18 years.
* Subject has a diagnosis of oral lichen planus deemed by the investigator to be of sufficient severity to require systemic agents. The diagnosis can be made by biopsy proven oral lichen planus or biopsy proven cutaneous lichen planus in the setting of a subject with oral disease consistent with lichen planus.
* Subject has a clinical lesion score of at least 2.
* If female of childbearing potential, subject will have a negative urine pregnancy test at screening and week 0.
* If female, subject will be either post-menopausal for > 1 year; surgically sterile (hysterectomy or bilateral tubal ligation); or practicing one form of birth control (abstinence, oral contraceptive, estrogen patch, implant contraception, injectable contraception, intrauterine device [IUD], diaphragm, condom, sponge, spermicides, or vasectomy of partner). Female subjects will continue to use contraception for 3 months following the last injection.
* Subjects must be on stable doses of topical medications, such as corticosteroids, cyclosporine, and tacrolimus for the past 4 weeks.

Exclusion Criteria:

* Patients with known hypersensitivity to Raptiva (efalizumab) or any of its components.
* Pregnant or lactating women
* Subject has evidence of a clinically significant, unstable or poorly controlled medical condition.
* Subject has a chest X-ray consistent with an active infection or previous exposure to tuberculosis (TB) and/or a positive purified protein derivative test at screening (> 5 mm). (Subjects may participate if they are being actively treated in accordance with Centers for Disease Control [CDC] guidelines.)
* Subject has a serious, active or recurrent bacterial, viral, or fungal infection. This includes hepatitis B and C, and HIV.
* Subject has been hospitalized for infection or received intravenous (IV) antibiotics within the previous 2 months prior to baseline.
* Subject has a history of tuberculosis without documented adequate therapy.
* Subject has been diagnosed with a malignancy within the past 5 years except for successfully treated non-melanoma skin cancer.
* Subject has any dermatologic disease in the target site that may be exacerbated by treatment or interfere with examination.
* Subject has been administered an investigational drug in another clinical study within 30 days prior to baseline (or 5 half-lives, whichever is longer). Subjects in observational studies without investigational drugs or devices may still be enrolled.
* Subject has used the following systemic agents within 4 weeks prior to week 0: photochemotherapy, systemic corticosteroids, cyclosporine, tacrolimus, azathioprine, methotrexate, mycophenolate mofetil, hydroxychloroquine, chloroquine, quinacrine, dapsone, or thalidomide.
* Subject has previously been treated with biologic immune response modifiers including alefacept, etanercept, infliximab, or adalimumab within 12 weeks prior to day 0 (or 5 half-lives, whichever is longer).
* Subject has previously been treated with efalizumab.
* Subject weighs over 125 kg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2005-01; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
primary efficacy measure will be oral mucosal surface area involvement | 12 weeks
  area of oral mucosa involvement was measured in cm2 at baseline, week 4, week 8, week 12 and week 20. the primary efficacy outcome measure was the change in oral mucosal involvement at week 12.

SECONDARY OUTCOMES:
clinical lesion score | Week 0, 1, 4, 8, 12, and 20
  a numerical score from 0 to 5 where 0 = no lesion; 1 = white striae only; 2 = white striae and erosion < 1 cm; 3 = white striae and erosion > 1 cm; 4 = white striae and ulceration < 1 cm; 5 = white striae and ulceration > 1 cm
ten centimeter visual analogue pain scale | Week 0, 1, 4, 8, 12, and 20
  Patients were asked to put an X on a 10 cm line that corresponded to their degree of pain where 0 cm represented no pain and 10 cm represented the most severe pain
oral health impact profile-14 questionnaire | Week 0, 1, 4, 8, 12, and 20
  The OHIP-14 is a validated measure of the negative impact of oral disease on an individual's well being. The impact of various oral problems are rated from "never" to "very often," which correlates to a score of 0 to 4. The responses are weighted and summated giving a maximum score of 56 and a minimum score of 0.
cutaneous surface area involvement | Week 0, 1, 4, 8, 12, and 20
  The area of cutaneous disease involvement was measured in cm2

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. Heffernan, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States